CLINICAL TRIAL: NCT05351320
Title: A Phase II Study of WX-0593 Combined With Concurrent Chemoradiotherapy in the Treatment of Unresectable Locally Advanced Non-small Cell Lung Cancer (NSCLC) With Activating Mutation of ALK or ROS1
Brief Title: WX-0593 Combined With Concurrent Chemoradiotherapy in Unresectable Locally Advanced NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jinming Yu (Other)
Responsible Party: Sponsor-Investigator, Jinming Yu, Director of the hospital, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FL006-IIT-002
Record Dates: First submitted 2022-04-24; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: NSCLC, Unresectable , Radiochemotherapy, WX-0593
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WX-0593 single arm (Experimental): Part 1: Participants will receive WX-0593 monotherapy until disease progression or unacceptable toxicity.
  Part 2: Participants will receive 1 or 2 cycles of WX-0593 monotherapy and subsequently with concurrent chemoradiation, followed by WX-0593 monotherapy until disease progression or unacceptable toxicity.
  Interventions: Drug: WX-0593 Tablets; Drug: chemotherapy; Radiation: Thoracic Radiation Therapy（TRT）

INTERVENTIONS:
Drug: WX-0593 Tablets — WX-0593 60 mg, tablets, orally, once daily for 7 days, followed by WX-0593 180 mg, tablets, orally, once daily
  Other Names: Iruplinalkib
Drug: chemotherapy — Platinum-based chemotherapy
Radiation: Thoracic Radiation Therapy（TRT） — Five days a week to accept chest radiotherapy, once per day, every time 1.8-2.0 Gy, total dose 54-66 Gy

SUMMARY:
The aim of this trial is to evaluate the safety of WX-0593 combined with concurrent chemoradiotherapy in unresectable, locally advanced non-small cell lung cancer (NSCLC) with activating mutation of ALK or ROS1. This trial consists of two parts. In Part 1, approximately 8 patients will be included and receive WX-0593 maintenance until disease progression or unacceptable toxicity. In Part 2, approximately 32 patients will be included and receive WX-0593 monotherapy for 1-2 cycles and subsequently with concurrent chemoradiation, followed by WX-0593 maintenance until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older;
* Pathologically confirmed NSCLC who present with investigator-assessed previously untreated, unresectable, locally advanced (Stage II、III) disease (according to TMN staging of AJCC version 8);
* Has active mutation of ALK or ROS1;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1;
* Has at least one evaluable lesion (according to RECIST 1.1);
* Have adequate pulmonary function test as a forced expiratory volume in 1 second (FEV1) >50% of predicted normal volume and carbon monoxide lung diffusing capacity (DLCO) >40% of predicted normal value;
* Have adequate organ and marrow function;
* If participant is a woman of childbearing potential (WOCBP), must agree to follow the contraceptive guidance from written informed consent until at least 180 days after the last dose of study treatment. The female participant should have negative serum pregnancy test within 7 days prior to the first dose of study drug, and not breastfeeding;
* A male participant must agree to use contraception from written informed consent until at least 180 days after the last dose of study treatment.

Exclusion Criteria:

* Diagnosed other malignant tumor besides NSCLC within 5 years prior to study entry;
* Mixed small cell and non-small cell lung cancer histology;
* Has received prior therapy with any ALK TKI;
* Has a history of extensive diffuse/bilateral interstitial fibrosis, or grade 3 or 4 pulmonary fibrosis or interstitial lung disease prior to the first dose of study drug.

Has a known history of active tuberculosis; severe infection within 4 weeks prior to study entry;

* History of primary immunodeficiency;
* Active or prior documented autoimmune disease within the past 2 years. NOTE: Patients with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Develop Grade 3 or Higher drug-related Pneumonitis | within 90 days after radiation therapy

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 24 months
  PFS is defined as the time from the first dose of study drug to the first documented disease progression or death due to any cause, whichever occurs first
Overall Survival (OS) | 24 months
  OS is defined as the time from the first dose of study drug to death due to any cause.
Adverse Events (AEs) | 24 months
  Percentage of participants who experienced one or more AEs.
Disease control rate (DCR) | 24 months
Objective response rate (ORR) | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China